CLINICAL TRIAL: NCT04799262
Title: Phase II Study of Efficacy and Safety of Tofacitinib in Patients With Polymyalgia Rheumatica
Brief Title: Tofacitinib as a GC Sparing Agent for Polymyalgia Rheumatica
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCs Sparing Regimen in PMR
Record Dates: First submitted 2021-03-04; First posted 2021-03-16 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-05

CONDITIONS: Polymyalgia Rheumatica; Effect of Drug; Safety Issues
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — tofacitinib; Prednisone

STUDY DESIGN:
Masking Description: Assessor and data analyst blindness. To avoid bias, physicians who assess disease activity will be blinded. Participants are required not to discuss their treatment regimen with physicians at each visit. The success of the blind method will be judged by requiring the assessors to determine the therapy of participants after each visit. When the database is locked, the statistician will carry on the data analysis in the hidden of therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tofacitinib+Prednisone (Experimental): Tofacitinib was given at the dose of 10mg daily through the 24 weeks. Prednisone (or equivalent oral GCs) of 15 mg daily at baseline willed be tapered to 2.5 mg or less within 20 weeks. Unless specifically considered by patients and physicians, the GC will be tapered followed the predefined taper regimen depending on the response to treatment judged by PMR-AS. The PMR-AS will be determined every two weeks; if<10 the GC daily dosage was decreased by 2.5mg; if>17, the GC daily dosage was increased to the previous dosage; if 10≤PMR-AS≤17, the GC daily dosage was maintained at the previous stable dose.
  Interventions: Drug: Tofacitinib 5 MG

INTERVENTIONS:
Drug: Tofacitinib 5 MG — Oral tofacitinib at the dose of 5mg twice a day was given for 24 weeks. Prednisone (or equivalent oral GCs) of 15 mg daily at baseline willed be tapered to 2.5 mg or less within 20 weeks. Unless specifically considered by patients and physicians, the GC will be tapered followed the predefined taper regimen depending on the response to treatment judged by PMR-AS. The PMR-AS will be determined every two weeks; if<10 the daily GC dosage was decreased by 2.5mg; if>17, the GC daily dosage was increased to the previous dosage; if 10≤PMR-AS≤17, the GC daily dosage was maintained at the previous stable dose.
  Other Names: Prednisone

SUMMARY:
Glucocorticoids are the cornerstone treatment for polymyalgia rheumatica but induce adverse events. The efficacy of the candidate drug Tofacitinib has not yet been demonstrated in controlled studies. The aim of the study is to investigate the efficacy and safety of Tofacitinib as a glucocorticoid sparing agent in patients with polymyalgia rheumatica.

DETAILED DESCRIPTION:
A two-stage, phase 2 clinical trial was conducted to test whether tofacitinib would take into effect as a glucocorticoid sparing agent in patients with polymyalgia rheumatica. Tofacitinib was given at the dose of 10mg daily through the 24 weeks. Patients were to receive prednisone in a dosage of 15mg daily (or equivalent oral GCs) at baseline and tapered to 2.5mg or less daily within 20 weeks. The primary endpoint was the response to treatment, defined as the achievement of sustained low disease activity (PMR-AS<7) with GC independence (prednisone≤2.5mg daily or equivalent oral GCs) for 4 weeks from week 20.

The trial will be conducted following a two-stage Simon minimax design. After 8 participants have completed their 24-week follow up there will be an interim analysis. If there are 3 or more failures out of these 8 then the trial will stop with the conclusion that the study of Tofacitinib should be abandoned. If there are fewer than 3 failures then the study will continue until a further 6 participants have received treatment, giving a total sample size of 14. If amongst these 14 participants there are 4 or more failures then it will be concluded that further study of Tofacitinib should be abandoned. If further study of the drug is not abandoned at either the interim of the final analysis, then a recommendation to conduct a comparative, randomized phase III trial will be made.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male between 50 and 85 years old.
2. PMR according to the ACR/ EULAR 2012 PMR classification criteria.
3. Patients must have erythrocyte sedimentation rate (ESR) ≥20 mm/hr and/or CRP ≥8 mg/L associated with highly active PMR (PMR-AS>17) within 2 weeks prior to screening.
4. Patient is willing and able to take prednisone of 15 mg/day at baseline.
5. Signed written informed consent.

Exclusion Criteria:

1. Presence of any other connective tissue disease, such as but not limited to giant-cell arteritis, systemic lupus erythematosus, systemic sclerosis, vasculitis, myositis, mixed connective tissue disease, and ankylosing spondylitis.
2. Concurrent diagnosis of active fibromyalgia, rhabdomyolysis or neuropathic muscular diseases.
3. Organ transplant recipient.
4. Any prior (within the defined period below) or concurrent use of immunosuppressive therapies but not limited to any of the following: ① Any prior use of tumor necrosis factor inhibitors, anti-IL-6 agents or JAK inhibitor; ② Alkylating agents including cyclophosphamide within 6 months of baseline; ③ Cell-depletion agents (e.g. anti-CD20) without evidence of recovery of B cells to baseline level; ④ Abatacept within 8 weeks of baseline; ⑤ Any prior use of csDMARDs at unstable dose for less than 12 weeks before baseline, e.g. cyclosporine, azathioprine, mycophenolate mofetil, leflunomide, MTX; ⑥ Concurrent use of systemic GCs for conditions other than PMR.
5. Evidence (as assessed by the investigators) of active infection, such as presence of hepatitis B surface antigen (HBsAg) or hepatitis C antibody in blood, human immunodeficiency virus (HIV) positivity.
6. Patients with a history of active or recurrent herpes zoster.
7. Patients who have had surgery within 4 weeks of screening or planned surgery during study.
8. Malignancy within 5 years prior to screening, except for non-melanoma skin cancer.
9. Pregnant or breastfeeding woman.
10. Any medical condition that could interfere with the implementation or interpretation of the study or with the safety of the patient during the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Response to treatment | 24 week
  Response to treatment is defined as the achievement of sustained low disease activity (PMR-AS<7) with GC independence (≤2.5mg/d) for 4 weeks from week 20

SECONDARY OUTCOMES:
Time till GC-free low disease activity within 24w | 24 week
  Time till GC-free low disease activity (PMR-AS<7) within 24 weeks
Time till first relapse within 24w | 24 week
  Time till first relapse (PMR-AS ≥7) within 24w
Cumulative GC dose at 24w | 24 week
  Cumulative glucocorticoids dose over time
Proportion of patients with sustained remission with GC independence for 4 weeks from week 20 | 24 week
  Proportion of patients with sustained remission (PMR-AS <1.5) with GC independence (≤2.5mg/d) for 4 weeks from week 20
Incidence of adverse events (AEs) and Serious AEs (SAEs) | 24 week
  Incidence of adverse events (AEs) and Serious AEs (SAEs) within 24 weeks
Change of disease activity by PMR-AS | 24 week
  Change of disease activity by PMR-AS within 24 weeks
Assessment of quality of life using the MHAQ | 24 week
  The Modified Health Assessment Questionnaire (MHAQ), reduced the number of items from 20 in the original HAQ to eight, and improved the feasibility in clinical practice when screening patients. The MHAQ score is calculated as the mean of the scores for each activity. Total score is between 0.0-3.0, in 0.125 increments. Higher scores indicate worse function and greater disability. MHAQ scores <0.3 are considered normal.
Assessment of quality of life using the EQ-5D | 24 week
  Health quality assessed by EuroQol five dimensions questionnaire. It is a preference-based measure that can be regarded as a continuous outcome scored on a -0.59 to 1.00 scale, with 1.00 indicating 'full health' and 0 representing dead.
Circulating serum cytokines, immunoregulators, and inflammatory parameters | 24 week
  On the circulating serum cytokines, immunoregulators (IL-6, IL-1, BLyS/BAFF, IL-6 receptor, gp130, etc.), B cells receptors, phenotype of circulating T- and B-cells will be collected at W0 and W24. On inflammatory parameters (CRP and ESR) every 4 weeks from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Li, MD, Study Chair — RenJi Hospital
Locations (1):
- Ren Ji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang L, Li J, Yin H, Chen D, Li Y, Gu L, Fu Y, Chen J, Chen Z, Yang S, Ye S, Li T, Lu L. Efficacy and safety of tofacitinib in patients with polymyalgia rheumatica: a phase 2 study. Ann Rheum Dis. 2023 May;82(5):722-724. doi: 10.1136/ard-2022-223562. Epub 2023 Jan 5. No abstract available. PMID 36604153